CLINICAL TRIAL: NCT00045188
Title: Phase II Trial of STI571 in Metastatic Breast Cancer
Brief Title: Imatinib Mesylate in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02491; IDO1-691; N01CM17003 (NIH); CDR0000256915 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate twice daily. Treatment continues for at least 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have metastatic breast cancer. Imatinib mesylate may stop the growth of cancer by blocking the enzymes necessary for tumor cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of STI571 in metastatic breast cancer (MBC) that demonstrates expression of CD117 (c-kit) and/ or PDGFR.

SECONDARY OBJECTIVES:

I. To determine the clinical activity of STI571 in MBC with expression of CD117 (ckit) and/ or PDGFR by evaluating progression-free survival (PFS).

II. To determine the toxicity profile and tolerability of STI571 in patients with MBC.

III. To define serum, tissue and imaging surrogate endpoints of activity of STI571 in MBC.

OUTLINE:

Patients receive oral imatinib mesylate twice daily. Treatment continues for at least 8 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic breast cancer
* Documented expression of CD117 (c-kit) or platelet-derived growth factor receptor

  * Adequate tumor tissue from either the primary tumor and/or metastatic disease available for evaluation
* Must have received prior chemotherapy with an anthracycline (doxorubicin or epirubicin) and/or taxane (paclitaxel or docetaxel) as adjuvant or for advanced disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Bone disease may not be only source of measurable disease
  * Pleural or peritoneal ascites are not considered measurable disease
* No known brain metastases
* Hormone receptor status:

  * Not specified
* Female or male
* Not specified
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST or ALT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No prior allergic reaction attributed to compounds of similar chemical or biologic composition to imatinib mesylate
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 1 week after study
* No concurrent biologic agents
* No more than 2 prior chemotherapy regimens for metastatic disease

  * Therapy with high-dose regimens or bone marrow transplantation considered 1 regimen
* At least 4 weeks since prior chemotherapy (6 weeks for carmustine or mitomycin) and recovered
* No concurrent chemotherapy
* Prior hormonal therapy for stage IV disease and/or as adjuvant therapy allowed
* At least 4 weeks since prior radiotherapy and recovered
* Prior localized radiotherapy that does not influence the signal of the evaluable lesion is allowed
* At least 2 weeks since prior minor surgery
* At least 4 weeks since prior major surgery
* Recovered from prior surgery
* Low-molecular weight heparin or heparin allowed for anticoagulation
* No concurrent warfarin
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent investigational therapies or agents
* No other concurrent anticancer therapy
* No concurrent intake of cola, orange juice, grapefruit, or orange or grapefruit sections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-08; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Objective tumor response (CR + PR), as determined by the RECIST criteria | Up to 2 years

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
Time to progression | Up to 2 years
  Reported using the Kaplan-Meier method with 95% confidence intervals indicated.
Overall survival | Up to 2 years
  Reported using the Kaplan-Meier method with 95% confidence intervals indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cristofanilli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States